CLINICAL TRIAL: NCT04548778
Title: Clinical Evaluation of BÜHLMANN Fecal Pancreatic Elastase (fPELA) Tests in the Diagnosis of Exocrine Pancreatic Insufficiency (PEI)
Brief Title: BÜHLMANN FPELA in the Diagnosis of Exocrine Pancreatic Insufficiency
Status: Completed | Type: Observational
Sponsor: Bühlmann Laboratories AG (Industry)
Responsible Party: Sponsor
Other Study IDs: fPELA_ClinPerform2020
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-08

CONDITIONS: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- exocrine pancreatic insufficiency (PEI): Established diagnosis of PEI based on a routine clinical diagnostic work-up including a treat-to-diagnose approach using Pancreatic Enzyme Replacement Therapy (PERT).
  Interventions: Diagnostic Test: BÜHLMANN fPELA assay
- no exocrine pancreatic insufficiency (no PEI): No evidence of PEI according to routine clinical diagnostic work-up including a treat-to-diagnose approach using Pancreatic Enzyme Replacement Therapy (PERT).
  Interventions: Diagnostic Test: BÜHLMANN fPELA assay

INTERVENTIONS:
Diagnostic Test: BÜHLMANN fPELA assay — BÜHLMANN fPELA assays are immunoassays for the quantitative determination of fecal pancreatic elastase in human stool samples.

SUMMARY:
The study shall determine the clinical performance of the BÜHLMANN fecal pancreatic elastase (fPELA) assays in the diagnosis of exocrine pancreatic insufficiency (PEI).

This is a observational and cross-sectional performance study. Specimens and clinical data are collected by a single study site.

Included are subjects for which pancreatic elastase testing was indicated due to a suspected exocrine pancreatic insufficiency and which were at least 18 years of age. Subjects which suffered from diarrhea (stool water content ≥ 75%) at the time of sample collection are excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* suspected exocrine pancreatic insufficiency
* at least 18 years of age.

Exclusion Criteria:

* diarrhea (stool water content ≥ 75%) at the time of sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included are subjects for which pancreatic elastase testing was indicated due to a suspected exocrine pancreatic insufficiency and which were at least 18 years of age. Following patient groups show an increased risk for developing an exocrine insufficiency: chronic pancreatitis, cystic fibrosis, diabetes, pancreatic resection. Eligible study subjects provide one stool sample which is forwarded to the study site within three days.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Clinical Performance of BÜHLMANN fPELA assays in the diagnosis of PEI | December 2021
  Diagnostic sensitivity and specificity of BÜHLMANN fPELA assays

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Rosendahl, MD, Principal Investigator — Universitätsklinikum der Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Universitätsklinikum Halle (Saale), Halle, Germany